CLINICAL TRIAL: NCT02367859
Title: A Pilot Study of Dabrafenib and Trametinib for Patients With BRAF Mutated Ameloblastoma
Brief Title: Dabrafenib and Trametinib in Treating Patients With BRAF Mutated Ameloblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, A. Dimitrios Colevas, Professor of Medicine (Oncology) and Otolaryngology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-32275; NCI-2015-00169 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ENT0043 (Other: OnCore)
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Ameloblastoma; BRAF Gene Mutation
Keywords: ameloblastoma; BRAF; odontogenic cancer; adamantinoma
MeSH Terms: conditions — Ameloblastoma; Adamantinoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (dabrafenib) (Experimental): Patients receive dabrafenib PO BID every 12 hours plus trametinib daily PO for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients whose disease is judged to be not amenable to resection will continue dabrafenib and trametinib indefinitely as long as there has not been tumor progression.
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Given PO
  Other Names: BRAF Inhibitor GSK2118436; GSK-2118436A; GSK2118436; Tafinlar
Drug: Trametinib — Given PO
  Other Names: Mekinist

SUMMARY:
This pilot clinical trial studies dabrafenib and trametinib in treating patients with ameloblastoma and a specific mutation (change) in the BRAF gene. Dabrafenib and trametinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To observe the response rate of ameloblastoma to dabrafenib and trametinib at 6 weeks.

SECONDARY OBJECTIVES:

I. Feasibility and safety in this patient population. II. Response will be assessed pathologically. III. Two main histologic assays for treatment response will be used: tumor necrosis and phosphorylated-mitogen-activated protein kinase kinase 1 (MEK), phosphorylated-extracellular signal-regulated kinase (ERK), and Ki-67 levels as measured by immunohistochemistry.

OUTLINE:

Patients receive dabrafenib orally (PO) twice daily (BID) every 12 hours and trametinib 2 mg daily PO for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients whose disease is judged to be not amenable to resection will continue dabrafenib and trametinib indefinitely as long as there has not been tumor progression.

After completion of study treatment, patients are followed up for at least 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of ameloblastoma; all stages are eligible; patients must have evaluable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* B-Raf proto-oncogene, serine/threonine kinase (BRAF) V600E or other known dabrafenib sensitive BRAF mutation in tumor by any Clinical Laboratory Improvement Amendments (CLIA) certified lab; may include, for example, Sanger sequencing, SNaPshot platform, immunohistochemistry, Foundation One tests, etc.)
* Life expectancy > 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Absolute neutrophil count (ANC) > 1.5 x10^9/L
* Platelet (PLT) > 99 x 10^9/L
* Hemoglobin > 8 g/dL
* Total bilirubin (Tbili) < 1.6 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) < 2.6 x ULN
* Alkaline phosphatase (alk phos) < 2.6 x ULN
* Serum creatinine < 1.6 x ULN or creatinine clearance > 50 ml/min
* Ability to understand and the willingness to sign a written informed consent document
* Patients of childbearing potential must agree to use effective contraception until at least 6 months after treatment with dabrafenib
* Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* Left ventricular ejection fraction equal to or greater than normal

Exclusion Criteria:

* No prior treatment with agents targeting BRAF mutant tyrosine kinases or radiation of target lesions
* Invasive malignancy other than ameloblastoma within 3 years, excluding curatively treated basal cell carcinoma, and other highly curable cancers such as early stage cutaneous squamous cell carcinoma (T1 NO) cervical carcinoma in situ (CIS), early stage prostate cancer, thyroid cancer or breast cancer
* Uncontrolled hypertension, chronic heart failure (CHF), or other major medical illness
* Prior allergic reactions attributed to compounds of similar chemical or biologic composition to dabrafenib
* Concomitant use of strong inhibitors (e.g., ketoconazole, nefazodone, clarithromycin, gemfibrozil) or strong inducers (e.g., rifampin, phenytoin, carbamazepine, phenobarbital, St John's wort) of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) or cytochrome P450, family 2, subfamily C, polypeptide 8 (CYP2C8)
* Concomitant use of proton pump inhibitors, H2-receptor antagonists, antacids
* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Pregnant or nursing patients; women of childbearing potential must have a negative pregnancy test within 14 days of enrollment
* Electrocardiogram (EKG) with QTcB (Bazett's formula) > 480 ms done within 14 days of enrollment
* Interstitial lung disease or pneumonitis
* A history of retinal vein occlusion (RVO)
* Congestive heart failure NYHA class III or worse (Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.)
* A history of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Colevas, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Stanford Cancer Institute Trials — http://cancer.stanford.edu/trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Dabrafenib): Patients receive dabrafenib orally twice daily every 12 hours plus trametinib daily orally for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients whose disease is judged to be not amenable to resection will continue dabrafenib and trametinib indefinitely as long as there has not been tumor progression.
Period: Overall Study
Arm/Group | Treatment (Dabrafenib)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Dabrafenib)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Tumor response was assessed per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Overall tumor response was assessed as the number of participants achieving either a complete response (CR) or a partial response (PR). The criteria are:
  * CR = Disappearance of all target lesions
  * PR = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Overall Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions, and/or the appearance of one or more new lesion(s)
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
  The outcome is reported as the number of participants achieving the different levels of tumor response per RECIST, a number without dispersion.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Dabrafenib)
Number analyzed (Participants) | 1
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Overall Response (OR) | 0
  Progressive disease (PD) | 0
  Stable disease (SD) | 1

2. Secondary Outcome: Percent Tumor Necrosis
Description: Percent of tumor necrosis at the time of endpoint biopsy or surgical resection will be assessed. The tumor specimen from resection will be examined and the volume of the necrosis compared to the volume of the total tumor determined by central pathology. Percent tumor necrosis, in increments of 10%, will be determined. The outcome will be reported as the mean percent tumor necrosis, with standard deviation.
Time Frame: 6 weeks
Population: On the basis of futility due to study closure with inadequate accrual, post-surgical research specimens were not analyzed.
Arm/Group | Treatment (Dabrafenib)
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Proliferation
Description: An immunohistochemical laboratory analysis to assess proliferation will be performed on the initial pre-treatment biopsy (baseline) vs either the endpoint tumor biopsy or the tumor specimen from the resection. Ki-67 immunohistochemistry will be scored by at least 2 pathologists using percentage positive cells as the primary metric. Proliferation will be assessed as the difference from baseline in Ki-67 labeling to the end of treatment (tumor biopsy or the tumor specimen). The outcome will be expressed as the mean, with standard deviation.
Time Frame: 6 weeks
Population: as for outcome 2
Arm/Group | Treatment (Dabrafenib)
Number analyzed (Participants) | 0

4. Secondary Outcome: Phosphorylation of Tumor Markers MEK and ERK
Description: An immunohistochemical laboratory analysis to assess phosphorylation of the tumor markers MEK and ERK on the initial pre-treatment biopsy (baseline) vs either the endpoint tumor biopsy or the tumor specimen from the resection. Immunohistochemistry will be scored by at least 2 pathologists using percentage positive cells and intensity of staining as the primary metrics. Phosphorylation of MEK and ERK will be assessed as the observed difference in phosphorylated MEK and ERK labeling from baseline to the end of treatment (tumor biopsy or the tumor specimen). The outcome will be expressed as the mean, with standard deviation.
Time Frame: 6 weeks
Population: as for outcome 2
Arm/Group | Treatment (Dabrafenib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Treatment (Dabrafenib)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Dabrafenib) (N=1)
Flu like symptoms (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Rash acneform (Skin and subcutaneous tissue disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dermatologic syndrome (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/59/NCT02367859/Prot_SAP_001.pdf